CLINICAL TRIAL: NCT06522893
Title: Comparison of Electrical Dry Needling and Therapeutic Exercise Versus Therapeutic Exercise in Patients With Nonspecific Chronic Neck Pain: A Randomized Clinical Trial
Brief Title: Electrical Dry Needling and Therapeutic Exercise Versus Therapeutic Exercise in Patients With Nonspecific Chronic Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP-0429-2023-C4-F2
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Dry Needling and Therapeutic exercise (Experimental): The group receiving dry needling combined with therapeutic exercise (n=35) will receive up to 6 sessions of stimulation at the active trigger points in the cervical region, according to Travell and Simons: occipitofrontalis, sternocleidomastoid, splenius capitis, anterior, middle, and posterior scalene muscles, upper, middle, and lower trapezius, and multifidus at the C6 level. Using ultrasound guidance, 0.25 mm x 25 mm needles will be inserted into the active. The needles will be connected to a TENS (transcutaneous electrical nerve stimulation) device (TensMed S82-Enraf Nonius), applying an asymmetric biphasic square wave current, low frequency (8 Hz), pulse duration of 250 μs, with an intensity perceived as mild to moderate, for 30 minutes. In addition, this group will undergo a protocol of specific therapeutic exercises for the cervical spine during the same electropuncture session and immediately afterward.
  Interventions: Other: Electrical Dry Needling and Therapeutic exercise
- Therapeutic Exercise (Active Comparator): The therapeutic exercise group (n=35) will perform progressive exercises for the cervical flexor and extensor muscles, once a week for 6 weeks (6 sessions in total, with each session lasting 30 minutes). The protocol includes activation and recruitment of the deep cervical flexor muscles, isometric co-contraction exercises for both deep and superficial flexors, and eccentric and isokinetic exercises for both flexors and extensors. Each week's session will include the exercises for that week, along with the exercises from previous weeks, as detailed in the specific cervical spine exercise table, which indicates sets, repetitions, contraction time, and rest periods.
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Other: Electrical Dry Needling and Therapeutic exercise — The group receiving dry needling combined with therapeutic exercise (n=35) will receive up to 6 sessions of stimulation at the active trigger points in the cervical region, according to Travell and Simons: occipitofrontalis, sternocleidomastoid, splenius capitis, anterior, middle, and posterior scalene muscles, upper, middle, and lower trapezius, and multifidus at the C6 level, bilaterally, once a week for 3 weeks. Using ultrasound guidance, 0.25 mm x 25 mm needles will be inserted into the active trigger points. The needles will be connected to a TENS (transcutaneous electrical nerve stimulation) device (TensMed S82-Enraf Nonius), applying an asymmetric biphasic square wave current, low frequency (2 Hz), pulse duration of 250 μs, for 30 minutes. In addition, this group will perform a protocol of specific therapeutic exercises for the cervical spine during the same electropuncture session and immediately afterward.
  Arms: Electrical Dry Needling and Therapeutic exercise
Other: Therapeutic exercise — The therapeutic exercise group (n=35) will perform progressive exercises for the cervical flexor and extensor muscles, once a week for 6 weeks (12 sessions in total). The protocol includes activation and recruitment of the deep cervical flexor muscles, isometric co-contraction exercises for both deep and superficial flexors, and eccentric and isokinetic exercises for both flexors and extensors. Each week's session will include the exercises for that week, along with the exercises from previous weeks, as detailed in the specific cervical spine exercise table, which indicates sets, repetitions, contraction time, and rest periods.
  Arms: Therapeutic Exercise

SUMMARY:
To compare the effectiveness of electrical dry needling combined with therapeutic exercise versus therapeutic exercise alone in patients with nonspecific chronic mechanical neck pain.

DETAILED DESCRIPTION:
Neck pain is highly prevalent, affecting 203 million people worldwide in 2020 and ranking eleventh in terms of years lived with disability. More than 50% of individuals will not recover from an acute episode and will experience recurrent neck pain within 1 to 5 years, leading to a persistent and chronic problem. Chronic neck pain can originate from a traumatic episode, such as whiplash, or it may not have a traumatic origin. In the latter case, in the absence of an identifiable pathoanatomic cause, it is classified as nonspecific chronic neck pain (NSNP). The GBD 2021 study acknowledges that the burden of neck pain has not been reduced in the past three decades and projects a significant increase in this absolute burden by 2050. Several studies have highlighted the urgency of prioritizing future research on preventing and treating this condition.

Clinical practice guidelines for the management of NSNP advocate for the use of exercise. Specifically, it has been shown that specific neck exercises are more effective than other types of alternative exercises in reducing pain and disability in patients with NSNP. In recent years, treatment based on electrical Dry Needling (DN) has gained popularity and has become an alternative to conventional treatment for soft tissue injuries, noted for its low incidence of significant side effects. This technique seeks to induce a local mechanical and microtraumatic response, optimizing the release of endogenous opioids, decreasing cortisol, improving microcirculation, and reducing proinflammatory mediators. All of this can contribute to improved motor control and pain relief. Additionally, the advent of ultrasound technology has provided new opportunities to improve the safety of this invasive approach.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 30 and 65 years with chronic cervical pain lasting 3 months or more and not receiving any other type of physiotherapy treatment.

Exclusion Criteria:

* Patients with sensory and/or coagulation disorders, history of spine surgery, cardiac complications, severe concurrent central or peripheral nervous system disease, epilepsy, needle phobia, disc pathology, or serious pathologies that may be the primary cause of chronic cervical pain (e.g., tumors, Arnold Chiari disease, vertigo syndrome, etc.) will be excluded, as they are contraindicated for transcutaneous electrical nerve stimulation (TENS).

Ages: 30 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Neck disability index | At baseline, at 6 weeks and at 2 months
  The neck disability index consists of 10 questions addressing functional activities such as personal care, lifting, reading, work, driving, sleeping, recreational, pain intensity, concentration and headache.

SECONDARY OUTCOMES:
Pain (Visual Analog Scale) | At baseline, at 6 weeks and at 2 months
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).
McGill Pain Questionnaire | At baseline, at 6 weeks and at 2 months
  The McGill Pain Questionnaire is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is a multi-dimesional tool for pain assessment and it has three components, which are the sensory intensity, the cognitive evaluation of pain and the emotional impact of pain.
Quality of Life (SF-36 quality of life questionnaire) | At baseline, at 6 weeks and at 2 months
  The SF-36 quality of life questionnaire assesses 8 domains including physical functioning, physical role, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
Quality of Sleep (Pittsburgh Quality of Sleep Questionnaire Index) | At baseline, at 6 weeks and at 2 months
  The Pittsburgh Quality of Sleep Questionnaire Index (PSQI) will be used to study the quality of sleep. It comprises 24 items where the subjects respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to the remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction.
Tampa scale for kinesiophobia | At baseline, at 6 weeks and at 2 months
  The 17-item Tampa scale for kinesiophobia assesses fear of movement or of injury or reinjury.
Pain Catastrophizing Scale | At baseline, at 6 weeks and at 2 months
  The Pain Catastrophizing Scale (PCS) is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. Catastrophizing is commonly described as an exaggerated negative orientation toward noxious stimuli and plays an important role in experiencing and coping with pain. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.
Treatment expectations | At baseline, at 6 weeks and at 2 months
  Questionnaire on treatment expectations and the patient's perception level
Expectations regarding cervical pain | At baseline, at 6 weeks and at 2 months
  Questionnaire on expectations regarding cervical pain
Cervical Range of Motion (Pro Motion Capture. Werium) | At baseline, at 6 weeks and at 2 months
  Cervical range of motion is assessed with the patient sitting comfortably on a chair, with both feet flat on the floor, hips and knees at 90º of flexion, and buttocks positioned against the back of the chair.
Active and Latent Myofascial Trigger Points (Number of trigger Points) | At baseline, at 6 weeks and at 2 months
  Myofascial Trigger Points will be explored in the following pairs of muscles: occipitofrontalis, splenius capitis, sternocleidomastoid, anterior scalene, middle scalene, posterior scalene, upper trapezius, middle trapezius, lower trapezius, supraspinatus, infraspinatus, and multifidus level C6.

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro Sánchez, Almería, Almeria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] GBD 2021 Neck Pain Collaborators. Global, regional, and national burden of neck pain, 1990-2020, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2024 Mar;6(3):e142-e155. doi: 10.1016/S2665-9913(23)00321-1. PMID 38383088
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Fandim JV, Nitzsche R, Michaleff ZA, Pena Costa LO, Saragiotto B. The contemporary management of neck pain in adults. Pain Manag. 2021 Jan;11(1):75-87. doi: 10.2217/pmt-2020-0046. Epub 2020 Nov 25. PMID 33234017
- [Background] Farrell SF, Smith AD, Hancock MJ, Webb AL, Sterling M. Cervical spine findings on MRI in people with neck pain compared with pain-free controls: A systematic review and meta-analysis. J Magn Reson Imaging. 2019 Jun;49(6):1638-1654. doi: 10.1002/jmri.26567. Epub 2019 Jan 5. PMID 30614121
- [Background] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Background] Verhagen AP. Physiotherapy management of neck pain. J Physiother. 2021 Jan;67(1):5-11. doi: 10.1016/j.jphys.2020.12.005. Epub 2020 Dec 24. No abstract available. PMID 33358545
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Parikh P, Santaguida P, Macdermid J, Gross A, Eshtiaghi A. Comparison of CPG's for the diagnosis, prognosis and management of non-specific neck pain: a systematic review. BMC Musculoskelet Disord. 2019 Feb 14;20(1):81. doi: 10.1186/s12891-019-2441-3. PMID 30764789
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Falla D, Jull G, Hodges P. Training the cervical muscles with prescribed motor tasks does not change muscle activation during a functional activity. Man Ther. 2008 Dec;13(6):507-12. doi: 10.1016/j.math.2007.07.001. Epub 2007 Aug 27. PMID 17720609
- [Background] Villanueva-Ruiz I, Falla D, Lascurain-Aguirrebena I. Effectiveness of Specific Neck Exercise for Nonspecific Neck Pain; Usefulness of Strategies for Patient Selection and Tailored Exercise-A Systematic Review With Meta-Analysis. Phys Ther. 2022 Feb 1;102(2):pzab259. doi: 10.1093/ptj/pzab259. PMID 34935963
- [Background] Fidalgo-Martin I, Ramos-Alvarez JJ, Murias-Lozano R, Rodriguez-Lopez ES. Effects of percutaneous neuromodulation in neuromusculoskeletal pathologies: A systematic review. Medicine (Baltimore). 2022 Oct 14;101(41):e31016. doi: 10.1097/MD.0000000000031016. PMID 36254060
- [Background] Romero-Morales C, Bravo-Aguilar M, Abuin-Porras V, Almazan-Polo J, Calvo-Lobo C, Martinez-Jimenez EM, Lopez-Lopez D, Navarro-Flores E. Current advances and novel research on minimal invasive techniques for musculoskeletal disorders. Dis Mon. 2021 Oct;67(10):101210. doi: 10.1016/j.disamonth.2021.101210. Epub 2021 Jun 4. PMID 34099238
- [Background] Rossi M, DeCarolis G, Liberatoscioli G, Iemma D, Nosella P, Nardi LF. A Novel Mini-invasive Approach to the Treatment of Neuropathic Pain: The PENS Study. Pain Physician. 2016 Jan;19(1):E121-8. PMID 26752480
- [Background] Chakravarthy K, Nava A, Christo PJ, Williams K. Review of Recent Advances in Peripheral Nerve Stimulation (PNS). Curr Pain Headache Rep. 2016 Nov;20(11):60. doi: 10.1007/s11916-016-0590-8. PMID 27671799
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816